CLINICAL TRIAL: NCT06379204
Title: A Study on the Intervention of Metabolic Syndrome Patients With Exercise Prescription Based on Ventilatory Threshold Using Cardiopulmonary Exercise Test
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taiyuan Central Hospital of Shanxi Medical University (Other)
Responsible Party: Principal Investigator, Liu Ruojiang, Chief Therapist, Taiyuan Central Hospital of Shanxi Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: No.2022026
Record Dates: First submitted 2024-04-18; First posted 2024-04-23 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Metabolic Syndrome X
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the maximum physiological value standardized group (Experimental)
  Interventions: Behavioral: the maximum physiological value standardized group
- the ventilatory threshold individualized group (Active Comparator)
  Interventions: Behavioral: the ventilatory threshold individualized group

INTERVENTIONS:
Behavioral: the maximum physiological value standardized group — 10 kcal/kg/week for 1-6 weeks, 12.5 kcal/kg/week for 7-12 weeks, exercise frequency of 3d/week, exercise intensity calculated by CPET measurement and HRR heart rate reserve method, gradually increasing.
  Arms: the maximum physiological value standardized group
Behavioral: the ventilatory threshold individualized group — 10 kcal/kg/week for 1-6 weeks, 12.5 kcal/kg/week for 7-12 weeks, exercise frequency of 3d/week, exercise intensity calculated by CPET measurement and three zone threshold model, gradually increasing.
  Arms: the ventilatory threshold individualized group

SUMMARY:
Analyze the clinical intervention effects and differences of progressive precision exercise prescriptions formulated by two methods for determining exercise intensity on metabolic syndrome (MS). Compare the effects of the two on the cardiovascular endurance of the MS population and verify the effectiveness of individualized methods in reducing absolute exercise intensity for MS patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients were included who met the Chinese Diabetic Society diagnostic criteria for MS-i.e., three or more of the following five items: (i) abdominal obesity (i.e., central obesity) with waist circumference ≥ 90 cm in males and ≥ 85 cm in females; (ii) hyperglycemia defined as fasting blood glucose ≥ 6.1 mmol/L or blood glucose ≥ 7.8 mmol/L two hours after glucose loading, or diagnosis of diabetes mellitus; (iii) hypertension defined as blood pressure ≥ 130/85 mmHg or diagnosed with hypertension; (iv) fasting triglycerides (TG) ≥ 1.70 mmol/L; and (v) fasting high-density lipoprotein cholesterol (HDL-C) < 1.04 mmol/L.
2. Patients were aged 25 to 65 years, with no restrictions on number of males or females.
3. Patients exhibited a long-term sedentary lifestyle and did not carry out moderate-intensity physical activity for at least three d/week of 30 min/d duration within three months of the study.
4. Patients were willing to participate and sign the informed consent form.

Exclusion Criteria:

1. Patients in an acute phase of various diseases or with organ failure, tumor, myocardial infarction, cardiac insufficiency, myocarditis, or chronic lung disease;
2. Patients with long-term alcohol consumption and those unable to ensure regular lifestyle habits during the intervention period;
3. Patients who were unable to ensure that they would carry out the stipulated exercise protocol during the intervention; and
4. Patients with drug modifications during the intervention that could affect the outcome markers.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2022-11-04 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-09-19 (Actual)

PRIMARY OUTCOMES:
Peak oxygen uptake | From enrollment to the end of 12 weeks of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Taiyuan Cardiac Rehabilitation Center, Taiyuan, Shanxi, China